CLINICAL TRIAL: NCT01796392
Title: Lung Function Improvement After Bronchoscopic Lung Volume Reduction With Pulmonx Endobronchial Valves Used in Treatment of Emphysema
Brief Title: Pulmonx Endobronchial Valves Used in Treatment of Emphysema (LIBERATE Study)
Acronym: LIBERATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 600-0012
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Emphysema
Keywords: emphysema; endobronchial valve; treatments; pulmonary rehabilitation; lung volume reduction
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBV and Optimal Medical Management (Experimental): This study arm will undergo EBV treatment along with optimal medical management, including smoking cessation program, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Interventions: Device: EBV
- Optimal Medical Management (Other): This study arm will receive maximal medical management, including smoking cessation program support if necessary, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Interventions: Other: Optimal Medical Management

INTERVENTIONS:
Device: EBV — This study arm will undergo EBV treatment and also receive optimal medical management, including smoking cessation program support, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Arms: EBV and Optimal Medical Management
Other: Optimal Medical Management — This study arm will receive optimal medical management, including smoking cessation program support, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  Arms: Optimal Medical Management

SUMMARY:
The purpose of this research is to study an investigational medical device that is designed to produce lung volume reduction in diseased areas of the lungs in patients with severe emphysema.

DETAILED DESCRIPTION:
The Pulmonx Zephyr Endobronchial Valve (EBV) is an implantable bronchial valve intended to decrease volume in targeted regions of the lung. It is indicated for the treatment of patients with severe emphysema. The EBV are placed in the diseased region of the lung using bronchoscopy. Bronchoscopy is a way to access the lungs using a small tube with a camera on the end. As the diseased region of the lung shrinks in size, healthier regions may expand and function more efficiently, resulting in improved breathing.

The LIBERATE Study is a clinical trial with two groups. Participants are assigned at random to the 'Treatment' group or to the 'Control' group. The 'Treatment' group will receive the Zephyr Endobronchial Valve (EBV) in combination with optimal medical therapy. The 'Control' group will receive optimal medical therapy alone. For every three participants in the study, two will go into the 'Treatment' group and one will go into the 'Control' group.

It is hypothesized that after placement of the EBV, lung function will be improved as compared to standard medical therapy alone.

Based on the 12-month follow up data from the LIBERATE Study, the Zephyr Endobronchial Valve System was approved by the FDA for the treatment of severe emphysema in June 2018. Following this PMA approval, and in agreement with the FDA, the ongoing long term follow-up (out to 5 years) of patients in the LIBERATE Study will now be conducted as a Post-approval study under the auspices of the "LIBERATE Extension Study". This is an administrative change with absolutely no change to the design or conduct of the study and, therefore has no material impact to the study participants or the study sites. All annual follow-up visits and evaluations are per the original LIBERATE Study protocol. Reporting to the FDA will be as the LIBERATE Extension Study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological evidence of emphysema
* Nonsmoking for 4 months prior to screening interview
* BMI less than 35 kg/m2
* Stable on current medication regimen
* Forced expiratory volume in one second (FEV1) between 15% and 45% of predicted value
* Residual Volume less than 175% predicted (determined by body plethysmography)
* Little or no collateral ventilation (CV-) as determined using the Chartis System

Exclusion Criteria:

* Had two or more hospitalizations over the last year for a COPD exacerbation
* Had two or more hospitalizations over the last year for pneumonia
* Had a prior lung transplant, lung volume reduction surgery, bullectomy or lobectomy
* Had a heart attack or congestive heart failure within the last 6 months
* Have heart arrhythmia
* Is alpha-1 antitrypsin deficient

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2023-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University Hospital, Philadelphia, PA
Locations (23):
- United States (17):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - University of California at Davis Medical Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Orlando Health, Orlando, Florida
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
- Brazil (2):
  - Hospital de Clinicas Porto Alegre, Porto Alegre, Rio Grande do Sul
  - INCOR - Hospital das Clinicas de Faculdade de Medicine da USP, São Paulo, São Paulo
- University Medical Center Groningen, Groningen, Netherlands
- United Kingdom (3):
  - Bristol Royal Infirmary, Bristol
  - University Hospital Llandough and University Hospital of Wales, Cardiff
  - Royal Brompton & Harefield NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bakker JT, Hartman JE, Klooster K, Charbonnier JP, Tsiaousis M, Vliegenthart R, Slebos DJ. Endobronchial valve treatment improves chest-CT diaphragm configuration in COPD. Respir Med. 2024 Nov-Dec;234:107856. doi: 10.1016/j.rmed.2024.107856. Epub 2024 Nov 6. PMID 39515624
- [Derived] Dransfield MT, Garner JL, Bhatt SP, Slebos DJ, Klooster K, Sciurba FC, Shah PL, Marchetti NT, Sue RD, Wright S, Rivas-Perez H, Wiese TA, Wahidi MM, Goulart de Oliveira H, Armstrong B, Radhakrishnan S, Shargill NS, Criner GJ; LIBERATE Study Group:. Effect of Zephyr Endobronchial Valves on Dyspnea, Activity Levels, and Quality of Life at One Year. Results from a Randomized Clinical Trial. Ann Am Thorac Soc. 2020 Jul;17(7):829-838. doi: 10.1513/AnnalsATS.201909-666OC. PMID 32223724
- [Derived] Criner GJ, Sue R, Wright S, Dransfield M, Rivas-Perez H, Wiese T, Sciurba FC, Shah PL, Wahidi MM, de Oliveira HG, Morrissey B, Cardoso PFG, Hays S, Majid A, Pastis N Jr, Kopas L, Vollenweider M, McFadden PM, Machuzak M, Hsia DW, Sung A, Jarad N, Kornaszewska M, Hazelrigg S, Krishna G, Armstrong B, Shargill NS, Slebos DJ; LIBERATE Study Group. A Multicenter Randomized Controlled Trial of Zephyr Endobronchial Valve Treatment in Heterogeneous Emphysema (LIBERATE). Am J Respir Crit Care Med. 2018 Nov 1;198(9):1151-1164. doi: 10.1164/rccm.201803-0590OC. PMID 29787288

RESULTS

PARTICIPANT FLOW:
Groups:
- EBV and Optimal Medical Management: This study arm will undergo The Zephyr Valve treatment along with optimal medical management, including smoking cessation program, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  EBV: This study arm will undergo EBV treatment and also receive optimal medical management, including smoking cessation program support, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
Period: Overall Study
Arm/Group | EBV and Optimal Medical Management | Optimal Medical Management
Started | 128 | 62
Completed | 119 (119 active subjects at 12-months) | 59 (59 active subjects at 12-months)
Not Completed | 9 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 5 | 1
Not completed — Excluded for medical reasons | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zephyr Valve Treatment and Optimal Medical Management: This study arm will undergo The Zephyr Valve treatment along with optimal medical management, including smoking cessation program, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
  EBV: This study arm will undergo Zephyr Valve treatment and also receive optimal medical management, including smoking cessation program support, pulmonary rehabilitation, usual medications and oxygen supplementation as necessary.
- Total: Total of all reporting groups
Arm/Group | Zephyr Valve Treatment and Optimal Medical Management | Optimal Medical Management | Total
Number analyzed (Participants) | 128 | 62 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.9) | 62.5 (7.1) | 63.5 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 29 | 101
  Male | 56 | 33 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 3 | 11
  White | 117 | 57 | 174
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 17 | 8 | 25
  United States | 88 | 42 | 130
  Brazil | 13 | 6 | 19
  United Kingdom | 10 | 6 | 16
Height [Mean (Standard Deviation); unit: inches] | 65.7 (4.0) | 66.3 (3.4) | 65.9 (3.9)
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.7 (3.9) | 24.3 (4.4) | 24.6 (4.1)
Pack Years Smoking History [Mean (Standard Deviation); unit: pack-years] — Calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  pack-years | 50.8 (26.9) | 48.6 (28.5) | 50.1 (27.4)
FEV1 Post-Bronchodilator (liters) [Mean (Standard Deviation); unit: liters] | 0.8 (0.3) | 0.8 (0.2) | 0.8 (0.2)
FEV1 Post-Bronchodilator (% predicted) [Mean (Standard Deviation); unit: %predicted] | 28.0 (7.5) | 26.2 (6.3) | 27.4 (7.1)
FVC (liters) [Mean (Standard Deviation); unit: liters] | 2.6 (0.9) | 2.6 (0.8) | 2.6 (0.8)
FVC (% predicted) [Mean (Standard Deviation); unit: %predicted] | 71.2 (16.0) | 68.5 (13.6) | 70.3 (15.3)
Diffusing Capacity (mL CO/min/mm Hg) [Mean (Standard Deviation); unit: mL CO / min / mmHg] — Population: Only 126 EBV subjects and 61 Control subjects were analyzed, due to missing data.
  mL CO / min / mmHg
    number analyzed (Participants) | 126 | 61 | 187
    (all) | 8.5 (3.5) | 8.3 (2.7) | 8.5 (3.2)
Diffusing Capacity (% predicted) [Mean (Standard Deviation); unit: %predicted] — Population: Only 126 EBV subjects and 61 Control subjects were analyzed, due to missing data.
  %predicted
    number analyzed (Participants) | 126 | 61 | 187
    (all) | 34.6 (11.3) | 33.1 (9.8) | 34.1 (10.9)
Residual Volume (RV) (liters) [Mean (Standard Deviation); unit: liters] — Population: Only 126 EBV subjects and 61 Control subjects were analyzed, due to missing data.
  liters
    number analyzed (Participants) | 126 | 61 | 187
    (all) | 4.7 (1.1) | 4.8 (0.9) | 4.7 (1.0)
Residual Volume (% predicted) [Mean (Standard Deviation); unit: %predicted] — Population: Only 126 EBV subjects and 61 Control subjects were analyzed, due to missing data.
  %predicted
    number analyzed (Participants) | 126 | 61 | 187
    (all) | 224.5 (42.5) | 224.6 (38.9) | 224.5 (41.2)
Total Lung Capacity (TLC) (liters) [Mean (Standard Deviation); unit: liters] — Population: Only 126 EBV subjects and 61 Control subjects were analyzed, due to missing data.
  liters
    number analyzed (Participants) | 126 | 61 | 187
    (all) | 7.5 (1.6) | 7.6 (1.4) | 7.6 (1.5)
Total Lung Capacity (% predicted) [Mean (Standard Deviation); unit: %predicted] — Population: Only 126 EBV subjects and 61 Control subjects were analyzed, due to missing data.
  %predicted
    number analyzed (Participants) | 126 | 61 | 187
    (all) | 133.5 (21.2) | 130.2 (12.4) | 132.4 (18.8)
GOLD Stage [Count of Participants; unit: Participants] — The GOLD system uses the term "stages" to refer to the different levels of COPD. Participants graded as GOLD Stage III are considered to have Severe COPD. Participants graded as GOLD Stage IV are considered to have Very Severe COPD.
  Participants
    GOLD Stage III | 54 | 16 | 70
    GOLD Stage IV | 74 | 46 | 120
6 Minute Walk Distance (m) [Mean (Standard Deviation); unit: meters] | 311.3 (81.3) | 301.9 (78.5) | 308.3 (80.3)
SGRQ Total score [Mean (Standard Deviation); unit: score on a scale] — The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations. Population: Only 127 EBV subjects and 61 Control subjects were analyzed, due to missing data.
  score on a scale
    number analyzed (Participants) | 127 | 61 | 188
    (all) | 55.2 (14.1) | 53.1 (14.1) | 54.5 (14.1)
mMRC Dyspnea Grade score [Mean (Standard Deviation); unit: score] — The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations. Population: Only 126 EBV subjects were analyzed, due to missing data.
  score
    number analyzed (Participants) | 126 | 62 | 188
    (all) | 2.4 (1.0) | 2.2 (0.8) | 2.4 (0.9)
BODE Index [Mean (Standard Deviation); unit: Index] — The BODE Index is comprised of a person's body mass index ("B"), airway obstruction ("O"), dyspnea ("D"), and exercise tolerance ("E"). Each of these components is graded on a scale of either 0 to 1 or 0 to 3. The final value-ranging from 0 to 10-provides doctors a percentage of how likely a person is to survive for four years. The final BODE tabulation is described as follows:
  0 to 2 points: 80 percent likelihood of survival 3 to 4 points: 67 percent likelihood of survival 5 of 6 points: 57 percent likelihood of survival 7 to 10 points: 18 percent likelihood of survival Population: Only 126 EBV subjects were analyzed, due to missing data.
  Index
    number analyzed (Participants) | 126 | 62 | 188
    (all) | 5.3 (1.5) | 5.3 (1.6) | 5.3 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1-second (FEV1)
Description: The percentage of study participants in the Zephyr Valve EBV (Endobronchial Valves) treatment arm meeting the clinically significant threshold of >15% improved forced expiratory volume in one second (FEV1), obtained immediately following bronchodilator therapy, as compared to the percentage in the control arm at 1 year post-procedure.
Time Frame: 1 year
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Zephyr Valve Treatment and Optimal Medical Management | Optimal Medical Management
Number analyzed (Participants) | 128 | 62
Participants | 61 | 10

2. Secondary Outcome: FEV1 Post-bronchodilator Absolute Change
Description: Difference between study arms in absolute change from baseline for post-bronchodilator FEV1 score at 1 year (value at 1 year minus value at baseline).
Time Frame: 1 year
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Zephyr Valve Treatment and Optimal Medical Management | Optimal Medical Management
Number analyzed (Participants) | 128 | 62
liters | 0.1 (0.2) | -0.003 (0.2)

3. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ)
Description: Difference between study arms in 'absolute change from baseline' for SGRQ score at 1 year (value at 1 year minus value at baseline).
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. The questionnaire comprises of two parts:
  Part I: Symptoms (frequency & severity) Part II: Activities that cause or are limited by breathlessness; Impacts (social functioning, psychological disturbances resulting from airways disease)
  A Total score is calculated which summarizes the impact of the disease on overall health status. Scores range from 0 to 100, with higher scores indicating more limitations.
Time Frame: 1 year
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zephyr Valve Treatment and Optimal Medical Management | Optimal Medical Management
Number analyzed (Participants) | 128 | 62
score on a scale | -7.6 (15.7) | -0.5 (15.5)

4. Secondary Outcome: 6-minute Walk Distance
Description: Difference between study arms in 'absolute and percentage change from baseline' for 6MWD at 1 year (value at 1 year minus value at baseline).
Time Frame: 1 year
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Zephyr Valve Treatment and Optimal Medical Management | Optimal Medical Management
Number analyzed (Participants) | 128 | 62
meters | 13.0 (81.5) | -26.3 (81.5)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Zephyr Valve Treatment and Optimal Medical Management | Optimal Medical Management
All-Cause Mortality (participants affected / at risk) | 5/128 | 1/62
Serious Adverse Events (participants affected / at risk) | 77/128 | 24/62
Other Adverse Events (participants affected / at risk) | 124/128 | 46/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zephyr Valve Treatment and Optimal Medical Management (N=128) | Optimal Medical Management (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Ulcer haemorrhage (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 5 (6)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 2 (2) | 0 (0)
Device expulsion (Product Issues) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 35 (50) | 21 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 40 (42) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zephyr Valve Treatment and Optimal Medical Management (N=128) | Optimal Medical Management (N=62)
Arrhythmia (Cardiac disorders) | 6 (7) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (9) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (11) | 0 (0)
Chest discomfort (General disorders) | 8 (8) | 0 (0)
Chest pain (General disorders) | 36 (46) | 1 (1)
Oedema peripheral (General disorders) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 7 (8) | 4 (4)
Infection (Infections and infestations) | 11 (12) | 5 (5)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 9 (10) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 11 (15) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 60 (99) | 25 (46)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (31) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (34) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT01796392/Prot_001.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT01796392/SAP_000.pdf